CLINICAL TRIAL: NCT03612674
Title: Adenoma Detection Rate With ARC Endocuff Vision Assisted Colonoscopy vs. Standard Colonoscopy in Colorectal Cancer Screening: a Multicenter Randomized Italian Study
Brief Title: Adenoma Detection Rate With Endocuff-Assisted Colonoscopy - an Italian Trial
Acronym: ITAvision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Prevention and Research Institute, Italy (Other)
Collaborators: Veneto Tumor Registry, Azienda Zero, Padua, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: F17G18000000007
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Colorectal Polyp; Colorectal Neoplasms
Keywords: Mass screening; Adenoma detection rate; ARC Endocuff Vision; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in two arms: a control-arm and an experimental-arm. Then arms data will be compared.
Who Masked: Participant
Masking Description: Participants will not be informed about diagnostic procedure in order to evaluate the acceptability of the exam with or without the studied device (in fact at the end of the examination care provider will ask participant about perceived pain during the procedure through the VAS score).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard colonoscopy (S) (Active Comparator): A standard colonoscopy will be performed.
  Interventions: Procedure: Standard colonoscopy
- AEV assisted colonoscopy (E) (Experimental): Colonoscopy with ARC Endocuff Vision attached to the top of the scope will be performed.
  Interventions: Device: ARC Endocuff Vision

INTERVENTIONS:
Procedure: Standard colonoscopy — Current standard of care colonoscopy.
  Arms: Standard colonoscopy (S)
Device: ARC Endocuff Vision — Subjects randomized to undergo a colonoscopy procedure with ARC Endocuff Vision will have this device placed on the top of the colonoscope used during their procedure.
  Arms: AEV assisted colonoscopy (E)

SUMMARY:
In European countries, colorectal cancer (CRC) represents an important public health problem. It is widely held view that most carcinomas develop from an adenoma-carcinoma progression.

Adenoma detection rate (ADR) is a marker of high quality colonoscopy and it was inversely associated with the risk of interval colorectal cancer, advanced-stage interval cancer, and fatal interval cancer after colonoscopy.

Although colonoscopy is considered the gold standard for adenoma detection, it has shown some limits, so industry has aimed at increasing detection rate of adenomas providing new technologies, most of witch to detect lesions located in blind spots.

ARC Endocuff Vision (AEV), the second generation of Endocuff, represents a new generation of these devices, thus assessing the diagnostic sensibility of ARC Endocuff Vision assisted colonoscopy (EAC) is an interesting challenge.

Aim of the study is to compare ADR of EAC versus standard colonoscopy among FIT positive subjects in the context of CRC screening programs.

DETAILED DESCRIPTION:
In European countries, colorectal cancer (CRC) represents an important public health problem. It is widely held view that most carcinomas develop from an adenoma-carcinoma progression.

It has been demonstrated that screening with fecal occult blood test (FOBT) significantly reduces mortality for CRC. Currently, population-based CRC screening programs using FOBT have been or are heading towards being implemented in many European countries. Fecal immunochemical test (FIT) has been adopted by most Italian Regions as the standard screening test, with total colonoscopy as diagnostic assessment in subjects resulted FIT positive. A significant impact of FIT-based screening on CRC mortality reduction has been observed in an Italian region after 10 years from screening implementation. Moreover, two studies carried out in a Northern-central area of Italy have shown a reduction in CRC incidence in subjects who attended FIT screening programs as compared to non-attendees.

Increasing colonoscopy quality is critical for the screening impact among population. Adenoma detection rate (ADR) is a marker of high quality colonoscopy and it was inversely associated with the risk of interval colorectal cancer, advanced-stage interval cancer, and fatal interval cancer after colonoscopy. ADR is defined as the proportion of colonoscopies during which at least one adenoma can be detected. A polish study showed that ADR was an independent predictor of the risk of interval colorectal cancer after screening colonoscopy. ADR has shown a direct correlation with: operator experience, cecal intubation, quality of bowel preparation, patient sedation, endoscope withdrawal time, presence of flat, depressed or subtle lesions, ability to visualize the proximal side of haustral folds, flexures (blind spots), rectal valves, and ileocecal valves.

On the other hand, colonoscopy is considered the gold standard for adenoma detection, but it has shown some limits. Data from colonoscopy studies showed that up to 25% of polyps were missed during colonoscopy and up to 8% of CRCs occurred within 3 years after a previous colonoscopy. Moreover, recent studies have shown that cancers post-colonoscopy are most likely due to missed lesions, rather than being new lesions.

For these reasons, industry has aimed at increasing detection rate of adenomas providing new technologies, most of witch to detect lesions located in blind spots.

ARC Endocuff Vision (AEV), the second generation of Endocuff, represents a new generation of these devices, thus assessing the diagnostic sensibility of ARC Endocuff Vision assisted colonoscopy (EAC) is an interesting challenge.

Previous researches have studied the performance of colonoscope distal attachment devices. More specifically, a 2016 meta-analysis of more than 5,000 patients demonstrates that, compared to traditional colonoscopy, the use of an Endocuff device improves ADR without any adverse effect on procedural efficiency or increased risk of significant adverse events. Moreover, Facciorusso et al. in 2017 assessed only a modest improvement in ADR by using distal attachment devices, especially in low-performing endoscopists, while in 2018 Williet showed, with moderate-quality evidence, an improvement in ADR with EAC without major adverse events, especially for operators with low-to-moderate ADR.

Second-generation AEV is a soft plastic cap, to be applied on the top of the colonoscopy. The cap has a propylene-made cylindrical core, with a single row of flexible arms. During the colon intubation procedure the device is nearly invisible, while in the retraction phase the arms begin to work, opening up and pulling the colon walls, stretching convoluted tracts.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a positive FIT result in the frame of national screening program

Exclusion Criteria:

* Subjects younger than 50 years old
* Active Inflammatory Bowel Disease
* Known condition of cholic stenosis
* Acute diverticulitis
* Patient not able to sign a informed consent form

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | Through study completion, an average of 1 year
  Comparison of the number of adenomas (ADR) detected per subject between the Endocuff Vision colonoscopy and the standard colonoscopy.

SECONDARY OUTCOMES:
Patient values | Day 1
  Comparison of ADR according to patient's age, sex, screening history (first or subsequent test) between the standard colonoscopy arm and the Endocuff Vision colonoscopy arm.
Exam values | Day 1
  Comparison of cecum intubation, patient discomfort (with Visual Analogue Scale -VAS) between the standard colonoscopy arm and the Endocuff Vision colonoscopy arm.
  The Visual Analogue Scale goes from 1 to 10, where 1 is the absence pain and 10 is severe pain.
  Number 1 represents the best outcome measure, while 10 is the worst result for this outcome measure.
Number of lesions | Day 1
  Comparison of polyps number between the standard colonoscopy arm and the Endocuff Vision colonoscopy arm.
Size | Day 1
  Comparison of polyps size between the standard colonoscopy arm and the Endocuff Vision colonoscopy arm.
Anatomical site | Day 1
  Comparison of polyps anatomical site between the standard colonoscopy arm and the Endocuff Vision colonoscopy arm.
Histological diagnoses | Through study completion, an average of 1 year
  Comparison of polyps histological diagnoses between the standard colonoscopy arm and the Endocuff Vision colonoscopy arm.
Colonoscopist' age | Through study completion, an average of 1 year
  Analysis of the involved colonoscopists' age.
Colonoscopist' years of experience | Through study completion, an average of 1 year
  Analysis of the involved colonoscopists' years of experience.
Colonoscopist' specialization | Through study completion, an average of 1 year
  Analysis of the involved colonoscopists' specialization.
Colonoscopist' number of exams in the previous year | Through study completion, an average of 1 year
  Analysis of the involved colonoscopists' number of exams in the previous year.
Colonoscopists' ADR in the previous year | Through study completion, an average of 1 year
  Analysis of the involved colonoscopists' ADR in the previous year.

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Amunni, MD, Study Director — Oncological Network, Prevention and Research Institute
Locations (12):
- Italy (12):
  - Santa Maria del Prato, Local Health Unit 1 Dolomiti, Veneto Region, Feltre, Belluno
  - San Martino Hospital, Local Health Unit 1 Dolomiti, Veneto Region, Belluno, BL
  - Maggiore Hospital, Crema Territorial Health Care Company, Lombardia Region, Crema, Cremona
  - Cazzavillan Hospital, Local Health Unit 8 Berica, Veneto Region, Arzignano, Vicenza
  - Screening Unit, Oncological Network, Prevention and Research Institute, Florence
  - San Paolo Hospital Company - University Campus, Milan
  - Sant'Antonio Hospital, Local Health Unit 6 Euganea, Veneto Region, Padua
  - Veneto Tumor Registry, Local Health Unit 4, Veneto Region, Padua
  - Santa Maria della Misericordia Hospital, Local Health Unit 5 Polesana, Veneto Region, Rovigo
  - Ca' Foncello Hospital, Local Health Unit 2 Marca Trevigiana, Veneto Region, Treviso
  - Molinette Hospital, Città della Salute e della Scienza University Hospital Company, Turin
  - San Bonifacio Hospital, Local Health Unit 9 Scaligera, Veneto Region, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zorzi M, Senore C, Da Re F, Barca A, Bonelli LA, Cannizzaro R, Fasoli R, Di Furia L, Di Giulio E, Mantellini P, Naldoni C, Sassatelli R, Rex D, Hassan C, Zappa M; Equipe Working Group. Quality of colonoscopy in an organised colorectal cancer screening programme with immunochemical faecal occult blood test: the EQuIPE study (Evaluating Quality Indicators of the Performance of Endoscopy). Gut. 2015 Sep;64(9):1389-96. doi: 10.1136/gutjnl-2014-307954. Epub 2014 Sep 16. PMID 25227521
- [Background] Giorgi Rossi P, Vicentini M, Sacchettini C, Di Felice E, Caroli S, Ferrari F, Mangone L, Pezzarossi A, Roncaglia F, Campari C, Sassatelli R, Sacchero R, Sereni G, Paterlini L, Zappa M. Impact of Screening Program on Incidence of Colorectal Cancer: A Cohort Study in Italy. Am J Gastroenterol. 2015 Sep;110(9):1359-66. doi: 10.1038/ajg.2015.240. Epub 2015 Aug 25. PMID 26303133
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Munroe CA, Lee P, Copland A, Wu KK, Kaltenbach T, Soetikno RM, Friedland S. A tandem colonoscopy study of adenoma miss rates during endoscopic training: a venture into uncharted territory. Gastrointest Endosc. 2012 Mar;75(3):561-7. doi: 10.1016/j.gie.2011.11.037. PMID 22341103
- [Background] Faiss S. The missed colorectal cancer problem. Dig Dis. 2011;29 Suppl 1:60-3. doi: 10.1159/000331119. Epub 2011 Nov 15. PMID 22104756
- [Background] Rees CJ, Rajasekhar PT, Rutter MD, Dekker E. Quality in colonoscopy: European perspectives and practice. Expert Rev Gastroenterol Hepatol. 2014 Jan;8(1):29-47. doi: 10.1586/17474124.2014.858599. Epub 2013 Dec 2. PMID 24410471
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Leufkens AM, van Oijen MG, Vleggaar FP, Siersema PD. Factors influencing the miss rate of polyps in a back-to-back colonoscopy study. Endoscopy. 2012 May;44(5):470-5. doi: 10.1055/s-0031-1291666. Epub 2012 Mar 22. PMID 22441756
- [Background] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Background] Pullens HJ, Siersema PD. Quality indicators for colonoscopy: Current insights and caveats. World J Gastrointest Endosc. 2014 Dec 16;6(12):571-83. doi: 10.4253/wjge.v6.i12.571. PMID 25512766
- [Background] le Clercq CM, Bouwens MW, Rondagh EJ, Bakker CM, Keulen ET, de Ridder RJ, Winkens B, Masclee AA, Sanduleanu S. Postcolonoscopy colorectal cancers are preventable: a population-based study. Gut. 2014 Jun;63(6):957-63. doi: 10.1136/gutjnl-2013-304880. Epub 2013 Jun 6. PMID 23744612
- [Background] Pohl H, Robertson DJ. Colorectal cancers detected after colonoscopy frequently result from missed lesions. Clin Gastroenterol Hepatol. 2010 Oct;8(10):858-64. doi: 10.1016/j.cgh.2010.06.028. Epub 2010 Jul 22. PMID 20655393
- [Background] Chin M, Karnes W, Jamal MM, Lee JG, Lee R, Samarasena J, Bechtold ML, Nguyen DL. Use of the Endocuff during routine colonoscopy examination improves adenoma detection: A meta-analysis. World J Gastroenterol. 2016 Nov 21;22(43):9642-9649. doi: 10.3748/wjg.v22.i43.9642. PMID 27920485
- [Background] Facciorusso A, Del Prete V, Buccino RV, Della Valle N, Nacchiero MC, Monica F, Cannizzaro R, Muscatiello N. Comparative Efficacy of Colonoscope Distal Attachment Devices in Increasing Rates of Adenoma Detection: A Network Meta-analysis. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1209-1219.e9. doi: 10.1016/j.cgh.2017.11.007. Epub 2017 Nov 11. PMID 29133257
- [Background] Williet N, Tournier Q, Vernet C, Dumas O, Rinaldi L, Roblin X, Phelip JM, Pioche M. Effect of Endocuff-assisted colonoscopy on adenoma detection rate: meta-analysis of randomized controlled trials. Endoscopy. 2018 Sep;50(9):846-860. doi: 10.1055/a-0577-3500. Epub 2018 Apr 26. PMID 29698990
- [Derived] Zorzi M, Hassan C, Battagello J, Antonelli G, Pantalena M, Bulighin G, Alicante S, Meggiato T, Rosa-Rizzotto E, Iacopini F, Luigiano C, Monica F, Arrigoni A, Germana B, Valiante F, Mallardi B, Senore C, Grazzini G, Mantellini P; ItaVision Working Group. Adenoma detection by Endocuff-assisted versus standard colonoscopy in an organized screening program: the "ItaVision" randomized controlled trial. Endoscopy. 2022 Feb;54(2):138-147. doi: 10.1055/a-1379-6868. Epub 2021 Apr 8. PMID 33524994
- Available data/document: Analytic Code — http://www.epiclin.it